CLINICAL TRIAL: NCT07120100
Title: Repetitive Transcranial Magnetic Stimulation for Chemotherapy-Induced Peripheral Neuropathy (CIPN) in Breast and Gynecologic Cancer Survivors: A Pilot Study
Brief Title: Transcranial Magnetic Stimulation for Chemotherapy-Induced Peripheral Neuropathy in Breast and Gynecologic Cancer Survivors
Acronym: rTMS for CIPN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI188734
Record Dates: First submitted 2025-07-30; First posted 2025-08-13 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer Female; Gynecologic Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Repetitive Transcranial Magnetic Stimulation (rTMS) Administration (Experimental)
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — Repetitive Transcranial Magnetic Stimulation will be administered Monday-Friday for two weeks (10 sessions total)

SUMMARY:
The goal of this study is to evaluate the change in pain scores among patients with chemotherapy-induced peripheral neuropathy after receiving treatment with repetitive transcranial magnetic stimulation (rTMS).

ELIGIBILITY:
Inclusion Criteria:

* Female subjects aged ≥ 18 years.
* Histologically confirmed breast or gynecologic cancer.
* Developed neuropathic pain with the initiation of or within one month after completion of treatment with anti-neoplastic agents from the following class:

  * Platinum-based drugs
  * Taxanes
  * Vinca alkaloids
* Pain score 4 or more on the Pain Numeric Rating Scale (PNRS).
* Score 3 or more on the Douleur Neuropathique 4 (DN-4) questionnaire.
* Persistent neuropathic pain with current use of at least one neuropathic medication.
* Subjects must have been on a stable dose of neuropathic pain medication for at least 6 weeks prior to enrollment.

  -- Note: Additional washout periods for other pain medications may be needed and will be determined by the Investigator.
* For female subjects: Negative pregnancy test or evidence of post-menopausal status. The post-menopausal status will be defined as having been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women < 50 years of age:

    * Amenorrheic for ≥ 12 months following cessation of exogenous hormonal treatments; and
    * Luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution; or
    * Underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
  * Women ≥ 50 years of age:

    * Amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments; or
    * Had radiation-induced menopause with last menses >1 year ago; or
    * Had chemotherapy-induced menopause with last menses >1 year ago; or
    * Underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy, or hysterectomy).
* Subjects of childbearing potential must agree to use a highly effective method of contraception as described in Section 5.4.1.
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

* Evidence of recurrent breast or gynecologic cancer at the time of enrollment.
* Current or planned treatment with chemotherapy.

  --Note: Other anti-cancer treatments (e.g. hormone therapy and targeted therapies) are allowed at the Investigator's discretion.
* History of seizure, epilepsy, or other conditions that would, in the opinion of the investigator, negatively impact the patient's safety or ability to participate in the study.
* Presence of neuropathic pain unrelated to systemic cancer therapy, including but not limited to: painful diabetic neuropathy, HIV-induced neuropathy, neuropathic pain from radiation therapy and underlying cancer/other medical conditions.
* Presence of implantable devices including spinal cord stimulators, dorsal root ganglion stimulators, deep brain stimulators, cochlear implants, intrathecal pain pumps, and intracranial metallic objects which are incompatible with rTMS administration in the opinion of the treating investigator.
* Subjects on medications that, in the opinion of the investigator, significantly lower seizure threshold will be excluded.
* Any condition that would, in the Investigator's judgment, contraindicate the subject's participation in the clinical study due to safety concerns or compliance with clinical study procedures.
* History of recent suicide attempt or active suicidal ideation that, in the opinion of the investigator, presents an increased risk for study participation
* Medical, psychiatric, cognitive, or other conditions that may compromise the subject's ability to understand the subject information, give informed consent, comply with the study protocol or complete the study.
* Enrollment in another study that, in the opinion of the investigator, would negatively impact study participation or cause undue burden for the subject.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 19 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2027-09-15 (Estimated); Study Completion 2028-09-15 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Numeric Rating Scale (PNRS) between screening and end of treatment in subjects who complete at least 7 rTMS treatments. | 5 months
  To assess the change in pain scores (0- no pain to 10-worst pain imaginable) after treatment with repetitive transcranial magnetic stimulation (rTMS) in patients with CIPN.

SECONDARY OUTCOMES:
The rTMS therapy will be considered safe if the proportion of subjects reporting treatment related grade 3 adverse device effects per Common Terminology Criteria for Adverse Events (CTCAE 5.0) is less than or equal to 5%. | 2 years
  To evaluate the safety of open-label 10-Hz rTMS of the motor cortex in individuals with CIPN.
The rTMS therapy will be feasible if at least 70% of the treated subjects can complete at least 70% of the treatment sessions. | 2 years
  To evaluate the feasibility of 10 sessions of open-label 10-Hz rTMS of the motor cortex in individuals with CIPN.
Change in Pain Numeric Rating Scale (PNRS) | up to 12 weeks after initiation of study intervention
  To evaluate the duration of pain (0- no pain to 10-worst pain imaginable) relief after treatment with rTMS.
Change in Patient-Reported Outcomes Measurement Information System - 29 items (PROMIS-29) v.2.1 | up to 12 weeks after initiation of the study intervention
  To evaluate the change in patient-reported outcomes.
  Each question usually has five response options ranging in value from one to five. The raw score is the sum of the values of the response to each question. From the raw score, the T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10.
  This outcome measure will report the mean T-scores of 8 subscales; Physical Function (Range: 22.5-57), Anxiety (40.3-81.6), Depression (41.0-79.4), Fatigue (33.7-75.8), Sleep Disturbance (32-73.3), Social Roles (27.5-64.2), Pain Interference (41.6-75.6), and Cognitive Function (29.5-61.2).
Change in Brief Pain Inventory-Short Form (BPI-SF) Scores | up to 12-week after initiation of the study intervention
  To evaluate the change in patient-reported outcomes. This outcome measure will report two BPI-SF subscales.
  Pain Severity Score is the mean of 4 items. Scores range from 0-10, with lower scores indicating less pain and higher scores indicating more pain.
  Pain Interference Score is the mean of 7 items. Scores range from 0-10, with lower scores indicating less pain interference and higher scores indicating more pain interference.
  This outcome measure will report the mean of the Pain Severity and Pain Interference Scores.
Change in Patient's Global Impression of Change (PGIC) Score | up to 12-week after initiation of the study intervention
  To evaluate the change in patient-reported outcomes.
  The PGIC asks patients to rate how their pain has changed since the start of the study. This outcome measure will report the mean of the single-item, 7-point PGIC scale from 0 No change (or the condition has gotten worse) to 7 A great deal better, and considerable improvement that has made all the difference.
Change in EuroQol 5-Dimension, 5-Level (EQ-5D-5L) | up to 12-week after initiation of the study intervention
  To evaluate the change in patient-reported outcomes.
  The EQ-5D-5L assesses health status across five dimensions: Mobility, Self-care, Usual Activities, Pain/Discomfort, and Anxiety/Depression. Each dimension is rated from Level 1 (no problems) to Level 5 (extreme problems).
  For analysis, each dimension will be dichotomized into two categories: No Problems (Level 1) Problems (Levels 2-5) The outcome measure will report the number of participants in each category for each health dimension.
Change in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Chemotherapy-Induced Peripheral Neuropathy 20 (EORTC-QLQ-CIPN-20) | up to 12-week after initiation of the study intervention
  To evaluate the change in patient-reported outcomes.
  The EORTC QLQ-CIPN20 is 20 items on a 1-4 Likert scale, where 1 is "not at all" and 4 is "very much". Items are summed to obtain the raw score, then converted to a 0-100 scale.
  Higher scores indicate more severe chemotherapy-induced peripheral neuropathy (CIPN), lower scores indicate less CIPN

CONTACTS AND LOCATIONS:
Locations (1):
- Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah, United States